CLINICAL TRIAL: NCT00924573
Title: Double-blinded Comparative Study to Investigate the Efficacy and Safety of HOE490 O (Glimepiride and Metformin) Compared With Placebo on Top of Glimepiride in Patients With T2DM Inadequately Treated With Constant Dose of Glimepiride
Brief Title: Comparative Study of HOE490 O (Glimepiride and Metformin) Compared With Placebo on Top of Glimepiride
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC10846; HOE490/4045
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glimepiride; Metformin; Combination Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Metformin on top of glimepiride
  Twice a day with 2-6 mg of daily dose for glimepiride and 500-750mg of daily dose for metformin for 24 weeks
  Interventions: Drug: Metformin; Drug: Glimepiride (HOE490)
- 2 (Placebo Comparator): Placebo on top of glimepiride
  Twice a day with 2-6 mg of daily dose for glimepiride and 2-3 tablets of placebo for 24 weeks
  Interventions: Drug: placebo; Drug: Glimepiride (HOE490)

INTERVENTIONS:
Drug: Metformin — oral administration
  Arms: 1
Drug: placebo — oral administration
  Arms: 2
Drug: Glimepiride (HOE490) — oral administration

SUMMARY:
Primary objective of this study is to confirm the efficacy of HOE490 O (glimepiride/metformin) compared with placebo on top of glimepiride in HbA1c change.

Secondary objectives of this study is to evaluate the safety of HOE490 O (glimepiride/metformin) compared with placebo on top of glimepiride as well as other efficacy parameters

DETAILED DESCRIPTION:
Patients treated with 2-6mg/day of glimepiride will be recruited. The study period consists of screening phase of 6 weeks and double-blinded phase of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus patients treated with constant dose of glimepiride on top of diet and exercise
* Patients who gave informed consent to participate in the study

Exclusion Criteria:

* Patients with HbA1c of < 7.0 % and > 11.0 %
* Patients with any following laboratory test abnormality :

  * ALT and/or AST: > 3 X ULN
  * Neutrophils: < 1,000/mm3 and/or platelets < 100,000/mm3
  * Hemoglobin: <11 g/dL
  * Creatinine: >= 1.3 mg/dL in case of male or >= 1.0 mg/dL in case of female

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c from baseline | 24 weeks

SECONDARY OUTCOMES:
Change in the ratio patients with < 7.0% of HbA1c | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kaku Kohei, Professor, Principal Investigator — Kawasaki Medical University
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan